CLINICAL TRIAL: NCT07116070
Title: Sarcopenia and Related Factors in Patients With Multiple Sclerosis
Status: Recruiting | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Mehmet Kaan ALTUNOK, Lecturer, Selcuk University
Other Study IDs: SelcukU_PT_MS_SARCOPENIA
Record Dates: First submitted 2025-07-24; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Multiple Sclerosis; Sarcopenia
Keywords: multiple sclerosis; sarcopenia; muscle strength; physical performance; nutrition
MeSH Terms: conditions — Multiple Sclerosis; Sarcopenia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- One group (Observational Cohort): MS patients (18 years and older) followed in the clinic.
  Interventions: Other: Clinical Assessments

INTERVENTIONS:
Other: Clinical Assessments — Participants will undergo the following assessments:
  * Muscle strength: Handgrip strength test (using a digital dynamometer),
  * Muscle mass: Bioelectrical impedance analysis (BIA) or DXA,
  * Physical performance: 6-minute walk test, 5-repetition sit-to-stand test,
  * Fatigue: Modified Fatigue Impact Scale (MFIS),
  * Disability: EDSS,
  * Nutritional status: Mini Nutritional Assessment (MNA),
  * Physical activity: Godin Leisure-Time Exercise Questionnaire,
  * Quality of life: MSQoL-54.

SUMMARY:
Multiple Sclerosis (MS) is a chronic disease affecting the central nervous system, exhibiting autoimmune and neurodegenerative properties. Neurological deficits, mobility limitations, and decreased muscle strength are commonly observed in MS patients as the disease progresses. The literature indicates that low physical activity levels and neurological deficits in individuals with MS can lead to decreased muscle mass and functional losses. Sarcopenia is a condition characterized by decreased skeletal muscle mass and strength associated with aging and chronic diseases, and studies on the prevalence of sarcopenia in MS patients are limited.

Recent studies have revealed a high prevalence of sarcopenia in MS patients, which can have negative effects on physical performance, quality of life, and disease progression. Low muscle mass in MS patients can accelerate the loss of motor function and increase the level of disability. Additionally, nutritional deficiencies and low protein intake seen in MS patients are among the factors that accelerate muscle loss.

Studies examining the relationship between MS and sarcopenia in the literature emphasize the importance of early diagnosis and intervention to improve patients' quality of life and functional independence. Factors such as muscle strength, physical activity level, and nutritional status should be assessed to determine the risk of sarcopenia in MS patients.

This study was designed to determine the prevalence of sarcopenia in patients with Multiple Sclerosis (MS) and to examine the relationship between sarcopenia and fatigue, disability level (EDSS), nutritional status, and physical activity level.

In this context:

* The prevalence of sarcopenia in MS patients will be determined,
* The relationship between sarcopenia and muscle strength, physical performance, and body composition will be evaluated,
* The effects of nutrition and physical activity on sarcopenia in MS patients will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older,
* Having been diagnosed with Multiple Sclerosis (confirmed by a neurologist),
* Being in a stable phase of the disease (having not had an attack in the last 3 months),
* Having preserved walking ability (EDSS score ≤6.5),
* Being able to give informed consent to participate in the study.

Exclusion Criteria:

* Having another neuromuscular disease.
* Having developed significant muscle loss within the last 6 months due to use of corticosteroids or immunosuppressive therapy.
* Having systemic diseases that can cause muscle loss, such as cancer, rheumatic diseases, or severe metabolic disorders.
* Having undergone major surgery or a history of serious trauma within the last 3 months.
* Being pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with MS who applied to the Selçuk University Faculty of Medicine Hospital MS Living Center
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
Body composition | Baseline
  Body mass and body composition will be measured with the help of Tanita brand device using bioelectrical impedance method. Information provided by the patient, such as height, age, gender, and physical activity level, is manually entered into the device. The device then transmits a very low level, harmless electrical current into the body and automatically analyzes body composition based on the transit time of this current. Parameters to be evaluated in body composition; body mass index (BMI = body mass: (kg)/height2 (m)2), fat mass expressed as a percentage of body mass (pFM), fat-free mass (FFM) expressed in kilograms and appendicular skeletal muscle mass (ASMM) and skeletal muscle mass (SMM) expressed in kilograms. The device automatically provides all the specified parameters during a single measurement. The measurements will be recorded on the previously prepared form.
Handgrip Strength | Baseline
  This will be used to assess muscle strength. The validity and reliability of this test has been previously established in the literature.
6-Minute Walk Test | 6 Minutes
  This will be administered to assess physical performance. This test has been shown to be valid and reliable in neurological disease populations.
Mini Nutritional Assessment Form (MNA) | Baseline
  This will be used to assess nutritional status.

SECONDARY OUTCOMES:
Demographic data and personal characteristics | Baseline
  Demographic information such as sociodemographic characteristics, medications used, comorbidities, education level, occupation, smoking, alcohol use, past medical history, and family history of the individuals included in the study will be recorded.
Godin Leisure Time Exercise Questionnaire | Baseline
  Will be applied to assess the level of physical activity.
Expanded Disability Status Scale (EDSS) | Baseline
  This will be administered by a neurologist to determine the level of disability in MS patients.
Modified Fatigue Impact Scale (MFIS) | Baseline
  This will be used to assess fatigue levels in MS patients. The validity and reliability of the Turkish version have been previously confirmed.
Multiple Sclerosis Quality of Life Scale-54 | Baseline
  This scale will be used to measure patients' quality of life. The MSQoL-54 scale is a tool specifically developed for MS patients.

CONTACTS AND LOCATIONS:
Overall Officials: İsmail ÖZSOY, Assoc. Prof. Dr., Principal Investigator — Selcuk University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Konya, Türkiye; Haluk GÜMÜŞ, Prof. Dr., Study Chair — Selçuk University, Faculty of Medicine, Department of Neurology, Konya, Türkiye; Gülşah ÖZSOY, Assist. Prof. Dr., Study Chair — Selcuk University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Konya, Türkiye; Zehra KORKUT, Assist. Prof. Dr., Study Chair — Selcuk University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Konya, Türkiye; Yasemin GEDİKLİ, Res. Asst., Study Chair — Selcuk University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Konya, Türkiye; Emel A ATAMAN AKTAŞ, Dr., Study Chair — Selçuk University, Faculty of Medicine, Department of Neurology, Konya, Türkiye; Omar E QUTOB, Dr., Study Chair — Selçuk University, Faculty of Medicine, Department of Neurology, Konya, Türkiye
Locations (1):
- Selcuk University Faculty of Medicine Hospital MS Life Center, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Background] Guigoz Y. The Mini Nutritional Assessment (MNA) review of the literature--What does it tell us? J Nutr Health Aging. 2006 Nov-Dec;10(6):466-85; discussion 485-7. PMID 17183419
- [Background] Vickrey BG, Hays RD, Harooni R, Myers LW, Ellison GW. A health-related quality of life measure for multiple sclerosis. Qual Life Res. 1995 Jun;4(3):187-206. doi: 10.1007/BF02260859. PMID 7613530
- [Background] Armutlu K, Korkmaz NC, Keser I, Sumbuloglu V, Akbiyik DI, Guney Z, Karabudak R. The validity and reliability of the Fatigue Severity Scale in Turkish multiple sclerosis patients. Int J Rehabil Res. 2007 Mar;30(1):81-5. doi: 10.1097/MRR.0b013e3280146ec4. PMID 17293726
- [Background] Kurtzke JF. Rating neurologic impairment in multiple sclerosis: an expanded disability status scale (EDSS). Neurology. 1983 Nov;33(11):1444-52. doi: 10.1212/wnl.33.11.1444. PMID 6685237
- [Background] Goldman MD, Marrie RA, Cohen JA. Evaluation of the six-minute walk in multiple sclerosis subjects and healthy controls. Mult Scler. 2008 Apr;14(3):383-90. doi: 10.1177/1352458507082607. Epub 2007 Oct 17. PMID 17942508
- [Background] Roberts HC, Denison HJ, Martin HJ, Patel HP, Syddall H, Cooper C, Sayer AA. A review of the measurement of grip strength in clinical and epidemiological studies: towards a standardised approach. Age Ageing. 2011 Jul;40(4):423-9. doi: 10.1093/ageing/afr051. Epub 2011 May 30. PMID 21624928
- [Background] Carvalho BM, Silva RSC, Lima VVM, Almondes KGS, Rodrigues FNS, D'Almeida JAC, Melo MLP. Excess weight increases the risk of sarcopenia in patients with multiple sclerosis. Mult Scler Relat Disord. 2023 Nov;79:105049. doi: 10.1016/j.msard.2023.105049. Epub 2023 Oct 8. PMID 37864991
- [Background] Gaemelke T, Pedersen IS, Dalgas U, Hvid LG. Sarcopenia in older people with multiple sclerosis: A cross-sectional study. Mult Scler Relat Disord. 2025 Jan;93:106190. doi: 10.1016/j.msard.2024.106190. Epub 2024 Nov 25. PMID 39631136
- [Background] Yuksel H, Balaban M, Tan OO, Mungan S. Sarcopenia in patients with multiple sclerosis. Mult Scler Relat Disord. 2022 Feb;58:103471. doi: 10.1016/j.msard.2021.103471. Epub 2021 Dec 26. PMID 34998245